CLINICAL TRIAL: NCT02198924
Title: A Study to Evaluate Efficacy and Safety of Postoperative Intravenous Parecoxib Sodium Followed by Oral Celecoxib Post Total Knee Arthroplasty in Osteoarthritis Patients
Brief Title: Efficacy and Safety of Postoperative Intravenous Parecoxib Sodium Followed by Oral Celecoxib in Osteoarthritis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Xisheng Weng, Department of Orthopedics, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WI1180091
Record Dates: First submitted 2013-07-17; First posted 2014-07-24 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Pain; Inflammation
Keywords: sequential administration; pain control; inflammation control; function recovery
MeSH Terms: conditions — Pain; Inflammation; Agnosia | interventions — parecoxib; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Parecoxib and Celecoxib (Experimental): Patients in the study group are supplied sequential treatment with Parecoxib 40 mg intravenously (IV) twice daily (Q12h) for the first 3 days post-surgery followed by Celecoxib 200mg orally twice daily (Q12h) up to 6 weeks post-surgery.
  Patient-controlled intravenous analgesia (PCIA) with Morphine is administrated to all the subjects starting immediately post-anesthesia and ending at 24h after operation. As long as oral intake is feasible, both the two groups may receive centrally-acting analgesic Tramadol Hydrochloride Sustained release tablets (TRAMCONTIN) as rescue analgesia if VAS score≧3.
  Interventions: Drug: Parecoxib and Celecoxib
- placebo (Placebo Comparator): Patients in the control group are supplied with the corresponding placebo with the same instructions.
  Patient-controlled intravenous analgesia (PCIA) with Morphine is administrated to all the subjects starting immediately post-anesthesia and ending at 24h after operation. As long as oral intake is feasible, both the two groups may receive centrally-acting analgesic TRAMCONTIN (Tramadol Hydrochloride Sustained release tablets) as rescue analgesia if VAS score≧3.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Parecoxib and Celecoxib — Patients in the study group are supplied sequential treatment with Parecoxib 40 mg intravenously (IV) twice daily (Q12h) for the first 3 days post-surgery followed by Celecoxib 200mg orally twice daily (Q12h) up to 6 weeks post-surgery.
  Arms: Parecoxib and Celecoxib
Drug: placebo — control patients are supplied with the corresponding placebo with the same instructions.
  Arms: placebo

SUMMARY:
In mainland China, knee Osteoarthritis (OA) is the leading cause of disability in older persons. Total knee arthroplasty (TKA) is now generally regarded by orthopaedic surgeons and patients as an effective treatment for end-stage knee OA in order to relieve pain, correct joint deformity and improve the life quality of patients.However, TKA has been called as one of the most painful Orthopedics surgery due to the weight bearing characteristics of knee joint and the high demand of functional exercise within the 6-8 weeks post operation. The targeted application of selective cyclooxygenase (COX) -2 inhibitor, such as Parecoxib or Celecoxib, can significantly reduce the level of inflammatory reaction one and two days postoperation . In addition, the perioperative administration of Celecoxib can directly or indirectly relieve postoperative pain, improve articular function and eventually augment life quality of the patients . Recently, effective treatment of post-operative pain with intravenous followed by oral COX-2 specific inhibitor has been demonstrated in many post-operative pain models . Significant morphine sparing effect and reduction of opioid distressed symptoms were also observed. In China, many surgeons have accept it as a routine strategy for controlling pain post TKA to sequentially give parecoxib 40 mg intravenously twice daily for the first 3 days post surgery and then Celecoxib 200mg orally twice daily. Although satisfactory results of this combination treatment on short-term pain reduction and functional improvement has been observed in clinical practice, high quality evidence is still lacking to prove its effect on the medium or long-term functionality recovery. This study is being conducted to investigate the combination regimen with intravenous parecoxib followed by oral celecoxib for post-surgical analgesic treatment in osteoarthritis patients undergoing total knee arthroplastic (TKA) surgery. Subjects will receive double-blinded study medication consisting of parecoxib injection in analgesic doses or matching placebo followed by oral celecoxib in acute pain doses or matching placebo in a double-blinded fashion. The hypothesis is subjects treated with parecoxib/celecoxib will consume less morphine over the first 24 hours of postoperation period, achieve improved pain control over study period, a quicker return to functionality, and has less opioid adverse events than those treated with opioids alone over 6-week recovery phase.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA), though generally regarded as an effective treatment for end-stage knee OA, has been called as "one of the most painful orthopedics surgeries" due to the weight bearing characteristics of knee joint and the high demand of functional exercise within the 6-8 weeks post operation.

Parecoxib and Celecoxib have been found to be able to relieve postoperative pain, spare opioid use, improve articular function and eventually augment life quality of the patients after TKA. In China, therefore, many surgeons have accept it as a routine strategy for controlling pain post TKA to sequentially use Parecoxib and then Celecoxib. However, high quality evidence is still lacking to prove its effect on the medium or long-term functionality recovery.

This multicenter, double blind, parallel-group randomized study, therefore, is aiming to evaluate efficacy and safety of postoperative intravenous Parecoxib sodium followed by oral Celecoxib in OA patients undergoing TKA. The hypothesis is that compared to placebo with opioids as rescue treatment, sequential use of Parecoxib/Celecoxib can achieve not only less morphine consumption over postoperatively 2 weeks, but also better pain control, quicker functional recovery, and less opioid related adverse events over 6-week recovery phase.

The primary objective of this study is to evaluate the morphine-sparing effects of the combination treatment with Parecoxib and Celecoxib versus placebo in subjects undergoing TKA. The secondary objective is to compare the effects of the combination treatment versus placebo on pain relief, inflammation control and functional rehabilitation after TKA. Total 86 subjects per group would have 90% power in detecting 100 mg or more in mean difference of morphine use on Day 14 between the two groups, assuming a common standard deviation of 200, and a two-sided alpha level of 0.05. This would result in a total 172 subjects. In consideration of 30% drop outs, 246 subjects would be adequate for the study. All subjects who meet the study inclusion and exclusion criteria will be randomly assigned in a 1:1 ratio to either Parecoxib/Celecoxib group or placebo group. The allocation or randomization will be study site based.Data will be collected using an Electronic Data Capture (EDC) under a strict intent-to-treat methodology, i.e., all the data of any Inform Consent Form signed subjects will be included in the study database.All subjects will be recruited from 4 study centers in China. The study will consist of 3 phases: an initial screening phase which must be completed within 30 days prior to randomization; a 6-week double blind treatment phase; and a 6 week follow up phase. A two-week wash-out procedure will be required before randomization for the patients with previous use of nonsteroidal antiinflammatory drug (NSAID) or COX-2 specific inhibitors.Variables considered continuous will be presented by descriptive statistics: number, mean, standard deviation, median, minimum, and maximum; and analyzed using parametric or non-parametric ANOVA, as appropriate. Variables considered categorical will be tabulated by frequency counts and percentages; and analyzed using Chi-square test or Fisher's exact tests. All the statistical tests will be two-sided with alpha=0.05, i.e., a p value <= 0.05 would be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is scheduled to undergo elective unilateral total knee arthroplasty because of OA, performed under a standardized regimen of general anesthesia, as specified in this protocol.
2. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
3. The subject is a male or female over 18 years of age.
4. Subjects of childbearing potential must agree to use an effective method of contraception throughout the study and for 42 days after the last dose of assigned treatment.
5. Total duration of the surgical procedure is four hours or less.
6. ASA grade 1-3 subjects.
7. Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, standardized rehabilitation scheme, and other study procedures.
8. The subject is in satisfactory health as determined by the investigator on the basis of medical history and physical exam.
9. The subject must demonstrate sufficient psychomotor dexterity and cognitive capacity to use intravenous (IV) patient-controlled analgesia(PCA).
10. The subject who live near to the hospital may be considered prior for the concern of convenient and sufficient follow-up.

    -

Exclusion Criteria:

1. The subject requires a revision to previous knee arthroplasty and/or is having a bilateral knee arthroplasties.
2. The subject requires an emergency knee arthroplasty.
3. Subject uses opioids more than three days/ week prior to operation unless they discontinue the opioids two months prior to screen.
4. Subject has a known hypersensitivity to COX-2 specific inhibitors, sulfonamides, lactose, NSAIDs, opioids or acetaminophen/paracetamol.
5. The subject has a history of arthritis:, chronic pain, metastasis, and Paget's disease.
6. The subject received any investigational medication within 30 days prior to the first dose of study medication.
7. The subject has any known laboratory abnormality, which in the opinion of the investigator, would contraindicate study participation ≧1.5 times the upper limit of the normal reference range.
8. The subject has an active malignancy of any type, or history of a malignancy (Subjects who have a history of basal cell carcinoma that has been successfully treated can be entered into the study.
9. Subject had any condition, which could preclude use of NSAIDs or COX-2 specific inhibitors.
10. The subject has active or suspected esophageal, gastric, pyloric channel, or duodenal ulceration history.
11. The subject has received warfarin or other anticoagulants during the 30 days preceding the first dose of study medication.
12. Subject is anticipated to require or requires treatment with lithium.
13. Subject is American Society of Anesthesiologists(ASA) grade 4-5.
14. The subject has a history of a psychiatric disorder requiring new or changing treatment
15. The subject has a history of uncontrolled chronic disease or a concurrent clinically significant illness, medical condition.
16. The subject has any cognitive impairment or other characteristics that would in the investigator's opinion preclude study participation or compliance with protocol mandated procedures.
17. Subject has a history of asthma or bronchospasm, which requires treatment with glucocorticoids.
18. Subject had a history of alcohol, analgesic or narcotic abuse.
19. Subject has been previously randomized into the study
20. Subjects who are investigational site staff members or relatives of those site staff
21. Participation in other studies within 3 months before the current study begins and/or during study participation
22. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation.
23. Pregnant females, breastfeeding females, or males and females of childbearing potential not using effective contraception.

    -

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Total narcotic use | Post-operative 2 WEEKS
  The sum of the cumulative Morphine consumption over the first 24 hours postsurgical period and the narcotic drug consumption till 72h, 2w post operation will be converted to morphine equivalents. The converting of tramadol to Morphine equivalents is estimated as 150mg Tramadol equals to 10mg of Morphine injection.

SECONDARY OUTCOMES:
Knee Society Score | post-operation 6 weeks
  For more than 20 years, The Knee Society's Knee Scoring System (KSS) has served as a simple, objective way to measure a patient's functional ability before and after total knee arthroplasty (TKA). KSS questionnaire generates three domain scores: KSS function score (walking, stairs and use of knee supports), range of motion and KSS score (pain, range of motion and stability) scores.
Western Ontario and McMaster Universities Arthritis(WOMAC) Index | prior to operation and at 2w,4w and 6w post operation
  The WOMAC is a widely used, proprietary set of standardized questionnaires to evaluate the condition of patients with knee osteoarthritis , including pain, stiffness, and physical functioning of the joints. A WOMAC test takes about 12 minutes, and is among the most widely used assessments in arthritis research.
Knee Society Score | prior to operation and at 2w and 4w post operation
  For more than 20 years, The Knee Society's Knee Scoring System (KSS) has served as a simple, objective way to measure a patient's functional ability before and after total knee arthroplasty (TKA). KSS questionnaire generates three domain scores: KSS function score (walking, stairs and use of knee supports), range of motion and KSS score (pain, range of motion and stability) scores.
Total Morphine use | over the first 24 hours postsurgical period
  The cumulative Morphine consumption over the first 24 hours postsurgical period.
Total narcotic use | 72h, 4w, 6w post operation
  The cumulative Morphine consumption and opioid drug over the first 24 hours postsurgical period.
Visual Analogue Scale | prior to operation and at 24h, 48h, 72h, 2w, 4w and 6w post operation
  A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured.
  Operationally a VAS is usually a horizontal line, 100 mm in length, anchored by word descriptors at each end. The patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined by measuring in millimetres from the left hand end of the line to the point that the patient marks.
EuroQol (EQ-5D) Score | prior to operation and 72h, 2w, 4w and 6w post operation
  EQ-5D is a standard instrument for use as a measure of health outcome. EQ-5D is primarily designed for self-completion by respondents and is ideally suited for use in postal surveys, in clinics and face-to-face interviews. It is cognitively simple, taking only a few minutes to complete. Instructions to respondents are included in the questionnaire.

OTHER OUTCOMES:
Knee circumference | prior to operation and at 72h, 2w, 4w and 6w post operation
skin temperature | prior to operation and at 72h, 2w, 4w and 6w post operation
Erythrocyte sedimentation rate(ESR) | prior to operation and at 72h, 2w, 4w and 6w post operation
C-Reactive Protein，CRP | prior to operation and at 72h, 2w, 4w and 6w post operation
interleukin-6 concentration in Synovial fluid | 0h, 24h and 48h post operation
interleukin-8 concentration in Synovial fluid | 0h, 24h and 48h post operation
interleukin-10 Synovial fluid concentration | 0h, 24h and 48h post operation
prostaglandin E2 concentration in Synovial fluid | 0h, 24h and 48h post operation
interleukin-6 concentration in Peripheral blood | prior to operation and at 72h, 2w, 4w and 6w post operation
interleukin-8 concentration in Peripheral blood | prior to operation and at 72h, 2w, 4w and 6w post operation
interleukin-10 concentration in Peripheral blood | prior to operation and at 72h, 2w, 4w and 6w post operation
prostaglandin E2 concentration in Peripheral blood | prior to operation and at 72h, 2w, 4w and 6w post operation
blood coagulation | prior to operation and at 72h, 2w, 4w and 6w post operation
The nature, incidence, duration, and severity of adverse events | until 6w post operation
Discontinuation due to adverse events | until 6w post operation
Adverse events | during and after trial medication discontinuation
complete blood count | 2 weeks post operation
blood chemistry parameters | 6w post operation
urinalysis test | 2 weeks post operation

CONTACTS AND LOCATIONS:
Overall Officials: Xisheng Weng, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carr AJ, Robertsson O, Graves S, Price AJ, Arden NK, Judge A, Beard DJ. Knee replacement. Lancet. 2012 Apr 7;379(9823):1331-40. doi: 10.1016/S0140-6736(11)60752-6. Epub 2012 Mar 6. PMID 22398175
- [Background] Du Q, Ge HJ, Zhu PF. Effects of perioperative analgesia on postoperative inflammatory response. Int J Anesth Resus., 2007, 28(1):48-53.
- [Background] Holm B, Kristensen MT, Bencke J, Husted H, Kehlet H, Bandholm T. Loss of knee-extension strength is related to knee swelling after total knee arthroplasty. Arch Phys Med Rehabil. 2010 Nov;91(11):1770-6. doi: 10.1016/j.apmr.2010.07.229. PMID 21044725
- [Background] Honsawek S, Deepaisarnsakul B, Tanavalee A, Sakdinakiattikoon M, Ngarmukos S, Preativatanyou K, Bumrungpanichthaworn P. Relationship of serum IL-6, C-reactive protein, erythrocyte sedimentation rate, and knee skin temperature after total knee arthroplasty: a prospective study. Int Orthop. 2011 Jan;35(1):31-5. doi: 10.1007/s00264-010-0973-0. Epub 2010 Feb 21. PMID 21203883
- [Background] Rasmussen GL, Steckner K, Hogue C, Torri S, Hubbard RC. Intravenous parecoxib sodium foracute pain after orthopedic knee surgery. Am J Orthop (Belle Mead NJ). 2002 Jun;31(6):336-43. PMID 12083587
- [Background] Hubbard RC, Naumann TM, Traylor L, Dhadda S. Parecoxib sodium has opioid-sparing effects in patients undergoing total knee arthroplasty under spinal anaesthesia. Br J Anaesth. 2003 Feb;90(2):166-72. doi: 10.1093/bja/aeg038. PMID 12538372
- [Background] Nussmeier NA, Whelton AA, Brown MT, Joshi GP, Langford RM, Singla NK, Boye ME, Verburg KM. Safety and efficacy of the cyclooxygenase-2 inhibitors parecoxib and valdecoxib after noncardiac surgery. Anesthesiology. 2006 Mar;104(3):518-26. doi: 10.1097/00000542-200603000-00020. PMID 16508400
- [Derived] Zhuang Q, Tao L, Lin J, Jin J, Qian W, Bian Y, Li Y, Dong Y, Peng H, Li Y, Fan Y, Wang W, Feng B, Gao N, Sun T, Lin J, Zhang M, Yan S, Shen B, Pei F, Weng X. Postoperative intravenous parecoxib sodium followed by oral celecoxib post total knee arthroplasty in osteoarthritis patients (PIPFORCE): a multicentre, double-blind, randomised, placebo-controlled trial. BMJ Open. 2020 Jan 9;10(1):e030501. doi: 10.1136/bmjopen-2019-030501. PMID 31924632
- [Derived] Zhuang Q, Bian Y, Wang W, Jiang J, Feng B, Sun T, Lin J, Zhang M, Yan S, Shen B, Pei F, Weng X. Efficacy and safety of Postoperative Intravenous Parecoxib sodium Followed by ORal CElecoxib (PIPFORCE) post-total knee arthroplasty in patients with osteoarthritis: a study protocol for a multicentre, double-blind, parallel-group trial. BMJ Open. 2016 Sep 8;6(9):e011732. doi: 10.1136/bmjopen-2016-011732. PMID 27609846